CLINICAL TRIAL: NCT00450606
Title: The Effects of Ambulatory Treatment at the Dead Sea on Osteoarthritis of the Knees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Collaborators: Lot Spa Hotel Dead Sea (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOR450007CTIL
Record Dates: First submitted 2007-03-21; First posted 2007-03-22 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Osteoarthritis of the Knees
MeSH Terms: interventions — Balneology; Hydrotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Balneotherapy and hydrotherapy

SUMMARY:
This study will check the efficacy of balneological therapy of bathing in Dead Sea fountain waters over a 6 week period on a twice a week basis (overall 12 treatments) in patients suffering from osteoarthritis of the knees.

DETAILED DESCRIPTION:
Since stay in the Dead Sea for a long period of time is an expensive matter, it is important to determine whether twice a week treatments can be as beneficiary as two straight weeks of treatments as was shown to be effective in previous studies.

Our study will follow the patients for a longer period of time (6 months) than was done in previous studies.

An additional advantage will be separating the therapeutical effect of our specific treatment from the therapeutical effect of being in a comfortable hotel away from the daily nuisances for 2 weeks which by itself has been shown to be pain relieving in patients suffering from rheumatic diseases.

Our study will take 50 patients suffering from Osteoarthritis of the knees and divide them in to 2 equal groups. One group will be treated twice a week with thermo-mineral baths at the temperature of 35-36 degrees Celsius for approximately 20 minutes. The other group will be treated twice a week with hot sweet water tub (without the water jets!) of the same temperature and for the same length of time.

Both groups will change nothing in their current medical treatment.

The patients will be examined at 5 points during this study: a few days before their first treatment, right after their last treatment (after 6 weeks), after one month, after 3 months and after 6 months.

All examination will be performed in the Soroka University Medical Center.

The clinical indexes and questionnaires which would be filled during this trial will be:

1. WOMAC index
2. Lequesne's index
3. Visual analogue scale by the patient
4. Visual analogue scale by the doctor
5. SF 36 and Health assessment questionnaire (HAQ)

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Osteoarthritis of the knees according to the conventional measurements of the American College of Rheumatology and who are treated in the Rheumatological clinics of the Soroka University Medical Center

Exclusion Criteria:

* Patients suffering from any other rheumatological disease other than osteoarthritis
* Patients that were previously treated with hydrotherapy or balneotherapy
* Patients suffering from balance disorders or loss of consciousness disorders such as epilepsy, arrhythmias etc.

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Quality of life evaluation at one, three and six months
Functional state of the patient at one, three and six months
Osteoarthritis severity at one, three and six months

CONTACTS AND LOCATIONS:
Overall Officials: Shaul Sukenik, Prof., Principal Investigator — Soroka University Medical Center